CLINICAL TRIAL: NCT03772366
Title: Genital Haemorrhage in Woman of Childbearing Age Treated for Venous Thromboembolism Disease : Comparison According to Oral Anticoagulant and Impact on Quality of Life.
Acronym: GENB-OAB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-17
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Genital Haemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Antivitamin K: Women in childbearing age treated for a venous thromboembolic disease with oral coagulant : Fluindione
- Rivaroxaban: Women in childbearing age treated for a venous thromboembolic disease with oral coagulant : Rivaroxaban
- Apixaban: Women in childbearing age treated for a venous thromboembolic disease with oral coagulant : Apixaban
- Control: Women in childbearing age with superficial venous insufficiency without treatment oral anticoagulant or antiplatelet.

SUMMARY:
Little data are available on the genital haemorrhages in woman of childbearing age treated for venous thromboembolic disease by oral anticoagulant, especially the impact on the quality of life. A recent systematic review in 2016 described for the first time in patients with venous thromboembolic a lower incidence in men of major haemorrhages and minor haemorrhages but clinically significant compared with women (5,3% and 7,9% respectively; RR: 0,635, 95%CI 0,54-0,74 ; p<0,001). It appears that this difference is related to genital haemorrhages and some direct oral anticoagulants are more associated with hemorrhagic surge. In post-hoc analyzes of phases III trials, rivaroxaban was most of the time associated with genital haemorrhages compared to vitamine K antagonists, effect not found with apixaban. Four other retrospective studies seem to find the same conclusions with a higher haemorrhagic risk with the rivaroxaban than with vitamine K antagonist or apixaban.

However, haemorrhagic risk is defined in these studies with criteria of severity (anemia, transfusion, use of a health professional, menstrual periods of more than 8 days, inter mentrual bleeding, presence of blood clots) and these studies do not take into account of minor haemorrhages that may affect on the quality of life and asthenia due to anemia.

Our objective is : 1- studying the proportion of women with abnormal genital haemorrhages among women of childbearing age treated for venous thromboembolism disease by oral anticoagulant including using a semi quantitative score of menorrhagia. 2- To compare this proportion according to the three molecules of oral anticoagulants (antivitamin K, rivaroxaban and apixaban) and compare the molecules two by two and 3- to evaluate the impact of these haemorrhages on the quality of life. Our study would have a control group of women of childbearing age followed in vascular medicine for superficial venous insufficiency without thrombosis and without oral anticoagulant because the proportion of genital haemorrhages in women of childbearing age in PACA region is not known.

ELIGIBILITY:
Inclusion Criteria E+ :

* Patient in childbearing age and >18 years
* Venous thromboembolic disease
* Oral anticoagulant treatment (fluindione, warfarine, rivaroxaban ou apixaban)
* Following by vascular doctor of Association Régionale des Médecins Vasculaires (ARMV) PACA (120 doctors) and/or one of the investigator center
* Affiliated with the Social Security Scheme
* Received an oral information

Inclusion Criteria E- :

* Patient in childbearing age and >18 years
* Superficial venous insufficiency
* No treatment with oral anticoagulant or anti platelet to not interfere with haemorrhage risk
* Following by vascular doctor of Association Régionale des Médecins Vasculaires (ARMV) PACA (120 doctors) and/or one of the investigator center
* Affiliated with the Social Security Scheme
* Received an oral information
* Non opposition register

Exclusion Criteria:

* <18 years patient
* Woman whose pregnancy is known
* Pre menopause
* Absence of menstruation
* Refusal to participate in the study
* No answer to the second call

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in childbaering age and major followed by a vascular doctor in Provence Alpes Côtes d'Azur region by one of the investigator centers or one of the 120 doctors in Association Régionale des Médecins Vasculaires ARMV PACA.
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of women with a major genital haemorrhage and/or a minor genital haemorrhage but clinically significant and/or a minor haemorrhage. | up to week 6
  Major genital haemorrhage : anemia (<12g/dl), transfusion ≥2 RBC (red blood concentrate) Clinically significant and/or a minor haemorrhage : FIGO recommendations (menstruation more than 8 days, inter menstrual bleeding, presence of blood clots, resort to health professionnal, dose or treatment modification Minor haemorrhage : semi-quantitated score Pictorial Blood Assessment Chart >100 (PBAC)

SECONDARY OUTCOMES:
Quality of life score measured with WHOQOL-BREF scale ( World Health Organization Quality of Life) | Day 1 and week 6
  WHOQOL-BREF scale comprises 26 items with 5 level of answer ("very poor" to "very good"), each answer give 4 scores 0 to 100 (higher scores = high level of quality of life) for the 4 domains following : physical health, mental health, social relationship and environment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier Arnaud, Study Director — Assistance Publique Hôpiaux Marseille
Locations (1):
- Assistance Publique Hôpitaux Marseille, Marseille, Bouches Du Rhônes, France